CLINICAL TRIAL: NCT07362771
Title: Effectiveness of Hatha Yoga With and Without Zumba Exercise on Clinical Outcomes in Females With Poly Cystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Latif Medical College (Other)
Responsible Party: Principal Investigator, Noor Fatima, House Officer Physical Therapy, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2024/169
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Poly Cystic Ovary Syndrome
Keywords: Anxiety; Poly-cystic ovarian syndrome; Females; Pain; Hatha Yoga
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Group A: Hatha Yoga With Zumba Exercise Patients received Zumba Exercise withHatha Yoga as baseline treatment. Group B: Hatha Yoga Patients received Hatha Yoga as baseline treatment.
Who Masked: Outcomes Assessor
Masking Description: The asessor was kept blind and was not aware of any intervetion groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zumba exercise (Experimental): Zumba exercises combine many sports steps that are easy to apply and help a person move many body muscles, such as arms, back, legs, and chest. Zumba exercises use physical strength, and all parts of the body are moved from head to toe. Zumba has a positive contribution to weight loss.This physical activity improves hormonal profile and reproductive function. In people undertaking physical activity regularly, under the influence of physical exercises, stress decreases, there is a lower increase in emotional tension.
  Interventions: Other: Hatha Yoga; Other: Zumba Exercise
- Hatha Yoga (Active Comparator): Hatha yoga is the most commonly practiced form of yoga in Western cultures - combines physical postures, mindful breathing, and meditation. Hatha yoga training comprised the following yoga poses: easy pose 1 min; breathing exercises 5 min; sun salutation 5 min; yoga relaxation 2 min; supported shoulder stand 1 min; fish pose 1 min; head knee pose 1 min; cobra 1 min; sitting half spinal twist 1 min; standing forward bend 1 min; extended triangle pose 1 min; yoga relaxation 5 min; breathing exercises 4 min; and easy pose 1 min.
  Interventions: Other: Hatha Yoga

INTERVENTIONS:
Other: Hatha Yoga — Hatha yoga is the most commonly practiced form of yoga in Western cultures - combines physical postures, mindful breathing, and meditation. Hatha yoga training comprised the following yoga poses: easy pose 1 min; breathing exercises 5 min; sun salutation 5 min; yoga relaxation 2 min; supported shoulder stand 1 min; fish pose 1 min; head knee pose 1 min; cobra 1 min; sitting half spinal twist 1 min; standing forward bend 1 min; extended triangle pose 1 min; yoga relaxation 5 min; breathing exercises 4 min; and easy pose 1 min.
Other: Zumba Exercise — Group A -Hatha Yoga with Zumba Exercise Group A was treated with Hatha Yoga and Zumba exercise for four weeks. Treatment was given by researcher himself.
  For Zumba exercise, patients were instructed to:
  (i) A warm up of 10 min with choreographies principally based on mobility, short displacements, and dynamic stretching (music from 125 to 135 bpm) (ii) A main part (40-45 min) based on the combination of different choreographies with Latin rhythms (merengue, salsa, reggae ton, music from 140 to 180 bpm) (iii) A final cool down (5-10 min) with choreographies based on soft Latin rhythms (salsa, music from 120-135 bpm) combined with breathing and stretching movements.
  (iv) All participants performed the Zumba Fitness sessions at the same time.(Barranco-Ruiz and Villa-González, 2020) Treatment frequency was two times a week. After four weeks treatment, the patient came for follow up at 6th week for final assessment.
  Arms: Zumba exercise

SUMMARY:
Effectiveness of Hatha Yoga with and without Zumba exercise on clinical outcomes in females with Poly Cystic Ovarian Syndrome-Randomized Clinical Trial

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine and metabolic disorder. PCOS is also one of the leading causes of infertility among women of reproductive age .Zumba are easy to apply and help a person move many body muscles, such as arms, back, legs, and chest. This includes aerobic exercise that can increase energy expenditure. Zumba exercises use physical strength, and all parts of the body are moved from head to toe. Zumba has a positive contribution to weight loss.Hatha yoga is combines physical postures, mindful breathing, and meditation. Yoga is most commonly practiced among adults who identify as female. Yoga can be practiced at home with minimal costs, making it potentially cost-effective and accessible to a wide audience.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged 23-28 year females ,hirsutism, irregular menses , anxiety,Pain,Poly Cystic Ovarian Syndrome Questionnaire,Medication.
* Pre-diagnosed cases of PCOS

Exclusion Criteria:

* Cardiovascular disease
* Endometrial cancer
* Diabetes mellitus
* Pregnancy
* Musculoskeletal injuries
* Hormonal contraceptives

Ages: 23 Years to 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females from age 23 to 28.
Enrollment: 54 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Pain Intenisty | Baseline and 4th week
  VAS used as clinical outcome tool for pain measurement.The visual analog scale (VAS) for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.

SECONDARY OUTCOMES:
Anxiety | Baseline and 4th week
  The Hamilton Anxiety Rating Scale (HAM-A) is a scale that measure the severity of anxiety in patients. The scale consists of 14 items designed to assess the severity of a patient's anxiety.

OTHER OUTCOMES:
PCOS symptoms | Baseline and 4th week
  The PCOS Questionnaire (PCOSQ) is a measurement tool for PCOS symptoms or its severity. It uses a 7-point scale to answer 26 questions in five domains: emotions, body hair, weight, infertility and menstrual problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data will be shared on request.

REFERENCES:
- [Background] Verma A, Upadhyay V, Saxena V. Effect of Yoga Therapy on Health Outcomes in Women With Polycystic Ovary Syndrome: A Systematic Review and Meta-Analysis. Am J Lifestyle Med. 2021 Aug 6;17(1):73-92. doi: 10.1177/15598276211029221. eCollection 2023 Jan-Feb. PMID 36636398
- [Background] ARGANA, G. A. M., CABAÑAS, K. P., CAJONTOY, M. K. P. C., MEDRANO, C. A. B. & PEREZ, C. J. G. THE EFFECT OF ZUMBA ON THE DISPOSITIONAL AFFECT OF SELECTED 3 RD YEAR CITE STUDENTS OF DLSL.